CLINICAL TRIAL: NCT05751876
Title: Clinical Experience of Dienogest in Perimenopausal Females With Symptomatic Adenomyosis
Brief Title: Dienogest in Perimenopausal Women With Adenomyosis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202207140RINB
Record Dates: First submitted 2023-02-13; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2022-07

CONDITIONS: Adenomyosis; Medication Adherence
Keywords: Adenomyosis; Perimenopause; Dienogest
MeSH Terms: conditions — Adenomyosis; Medication Adherence | interventions — dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with adenomyosis under dienogest: Perimenopausal women with symptomatic adenomyosis receiving dienogest
  Interventions: Drug: Dienogest

INTERVENTIONS:
Drug: Dienogest — Dienogest 2mg was prescribed once per day orally
  Other Names: Visanne, Bayer

SUMMARY:
Between September 2018 and December 2021, women who did not want further childbearing and received dienogest treatment for dysmenorrhea and/or hypermenorrhea were included in a retrospective chart review. Dienogest 2mg was prescribed once per day orally after completing the above-mentioned exam. The patient would return to our clinic on the 1st, 3rd, and 6th then every 3 months for a prescription. The primary outcome was successfully long-term (more than a year) dienogest use for pain and/or bleeding control. The secondary outcomes were the reasons for discontinuing dienogest treatment and the predictor of successful long-term treatment.

DETAILED DESCRIPTION:
Between September 2018 and December 2021, women who did not want further childbearing and received dienogest treatment for dysmenorrhea and/or hypermenorrhea were included in a retrospective chart review. The baseline demographic data included age, parity, delivery mode, and body mass index. Sonographic findings of adenomyosis, uterine size, and other gynecological lesions were recorded. Indications for dienogest treatment were analyzed, and women for pre-operative control or post-operative prevention of endometrioma were excluded. Women who were younger than 40 years old, with a post-treatment follow-up duration of fewer than 6 months, and medical conditions not suitable for dienogest treatment, such as known breast cancer, high thromboembolic effect, and smoking, were also excluded. The patients were further allocated into a younger group (more or equal to 40 years old and less than 45 years old) and an older group (more or equal to 45 years old to menopause).

For women with symptomatic adenomyosis, the pain scales and pretreatment data, including hormonal status, complete blood cell counts, liver function tests, and cancer antigen 125 (CA-125) as an indicator of endometriosis were recorded. Previous conservative treatment for adenomyosis was also reviewed. Dienogest 2mg was prescribed once per day orally after completing the above-mentioned exam. The patient would return to our clinic on the 1st, 3rd, and 6th then every 3 months for a prescription. During the treatment, blood tests and pelvic sonography would be performed every 6 months. Besides, a personal interview was also done for treatment effect evaluation and adverse effect management. Once the patient decided to discontinue the treatment, the follow-up started. The post-treatment follow-up interval was defined as the time frame between the day she stopped the dienogest treatment and her last visit on the medical record. The follow-up would include clinical symptoms of adenomyosis and laboratory or sonographic data if necessary. Menopause was defined when the FSH level was more than 30 mIU/mL with menopausal symptoms, such as hot flush, and no menstrual bleeding after stopping dienogest for a year.

The primary outcome was successfully long-term (more than a year) dienogest use for pain and/or bleeding control. The secondary outcomes were the reasons for discontinuing dienogest treatment and the predictor of successful long-term treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women with adenomyosis who did not want further childbearing and received dienogest treatment for dysmenorrhea and/or hypermenorrhea

Exclusion Criteria:

* < 40 y/o
* Post-operative prevention of endometriosis recurrence
* Medical conditions not suitable for dienogest treatment, such as known breast cancer, high thromboembolic effect, and smoking

Ages: 40 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with adenomyosis who did not want further childbearing and received dienogest treatment for dysmenorrhea and/or hypermenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
1 year dienogest use | September 2018 and December 2021
  successfully long-term (more than a year) dienogest use

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Hau Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The datasets analyzed during the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Result] Chiu CC, Hsu TF, Jiang LY, Chan IS, Shih YC, Chang YH, Wang PH, Chen YJ. Maintenance Therapy for Preventing Endometrioma Recurrence after Endometriosis Resection Surgery - A Systematic Review and Network Meta-analysis. J Minim Invasive Gynecol. 2022 May;29(5):602-612. doi: 10.1016/j.jmig.2021.11.024. Epub 2022 Feb 2. PMID 35123042
- [Result] Nirgianakis K, Vaineau C, Agliati L, McKinnon B, Gasparri ML, Mueller MD. Risk factors for non-response and discontinuation of Dienogest in endometriosis patients: A cohort study. Acta Obstet Gynecol Scand. 2021 Jan;100(1):30-40. doi: 10.1111/aogs.13969. Epub 2020 Sep 18. PMID 32767677
- [Result] Ono N, Asano R, Nagai K, Sugo Y, Nakamura T, Miyagi E. Evaluating the safety of dienogest in women with adenomyosis: A retrospective analysis. J Obstet Gynaecol Res. 2021 Apr;47(4):1433-1440. doi: 10.1111/jog.14612. Epub 2021 Feb 15. PMID 33590656
- [Result] Miyagawa C, Murakami K, Tobiume T, Nonogaki T, Matsumura N. Characterization of patients that can continue conservative treatment for adenomyosis. BMC Womens Health. 2021 Dec 28;21(1):431. doi: 10.1186/s12905-021-01577-x. PMID 34961515
- [Result] Neriishi K, Hirata T, Fukuda S, Izumi G, Nakazawa A, Yamamoto N, Harada M, Hirota Y, Koga K, Wada-Hiraike O, Fujii T, Osuga Y. Long-term dienogest administration in patients with symptomatic adenomyosis. J Obstet Gynaecol Res. 2018 Aug;44(8):1439-1444. doi: 10.1111/jog.13674. Epub 2018 May 29. PMID 29845696